CLINICAL TRIAL: NCT01078506
Title: Prevalence of Intracranial Aneurysm in Hong Kong Chinese
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, George KC Wong, Professor (Clinical), Chinese University of Hong Kong
Other Study IDs: GW006
Record Dates: First submitted 2010-02-26; First posted 2010-03-02 (Estimated); Last update posted 2013-04-23 (Estimated); Status verified 2013-04

CONDITIONS: Intracranial Aneurysm
Keywords: Chinese; intracranial aneurysm; magnetic resonance imaging
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Hong Kong Chinese: Without a history of known intracranial pathologies.

SUMMARY:
Intracranial aneurysm (localized dilatation in weakened blood vessel wall) rupture is a catastrophic disease, with half of the victims died and many of the survivors disabled. There is currently no data in the literature for the Chinese population concerning the prevalence, characteristics (location and size) and risk of harboring an unruptured intracranial aneurysm. In this study, the investigators aim to study the population prevalence and characteristics (location and size) of intracranial aneurysm in Hong Kong Chinese, and its cost-effectiveness. The screening is carried out using magnetic resonance angiography (MRA), with a 3-T magnetic resonance system, which is a well-established non-invasive method for intracranial aneurysm detection.

DETAILED DESCRIPTION:
As charted below.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged between 21 and 65 years

Exclusion Criteria:

* Contraindications to MRI
* History of known intracranial pathologies

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hong Kong Chinese without a history of known intracranial pathologies
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2010-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Intracranial aneurysm | Three years

SECONDARY OUTCOMES:
Other intracranial pathologies | Three years

CONTACTS AND LOCATIONS:
Overall Officials: George KC Wong, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Department of Surgery, The Chinese University of Hong Kong, Hong Kong, China